CLINICAL TRIAL: NCT06647381
Title: Implant-related Outcomes in the Context of Maxillary Sinus Lifting: A Prospective Study With 25 Years Follow-up
Brief Title: Implant-related Outcomes in the Context of Maxillary Sinus Lifting
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01280
Record Dates: First submitted 2024-10-03; First posted 2024-10-17 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Dental Implants
Keywords: Dental Implants; Sinus lift

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sinus lifting: Patients from a previous cohort of patients that received dental implants with sinus augmentation procedures

SUMMARY:
The population of interest will be recruited out of a cohort of patients who were initially treated at the Department of Oral Surgery and Stomatology between 1997 and 2001. The findings from a total of 56 patients that received tooth replacement treatment with dental implants during this period, were previously published in 2008. Now, 20 years later, the investigators will potentially recruit and re-examine as many patients as possible out of this original cohort. Exclusion criteria will be patients not able to come to the re-examination, concomitant diseases that compromise the health of this subject during the comprehensive examination (i.e., active severe infectious diseases, liver or kidney dysfunction/failure, currently under treatment), pregnant women, or unwilling to sign the consent form. Besides them, no further exclusion criteria are defined as patients receiving no intervention. The investigators assume that will be able to retrieve 40 patients having roughly 80 implants with sinus floor augmentation.

Recruitment, screening, and informed consent procedure

Patients treated at the Department of Oral Surgery between 1997 and 2001 and who were included in the previous case series study will be potentially recruited. Patients who are willing to participate will receive informed consent. The risks and benefits of being part of this study will be thoroughly explained to the patients without a limit of time. All the questions will be answered. After signing the informed consent patients will be examined. The participants will not be charged any costs for the recall examination.

Study procedures

After ethical approval, available patients will be screened and recruited for a re-examination visit. The anamnesis of the patients will be assessed using a questionnaire. In case of uncertainties regarding the medical history, a report from the patient's physician will be requested. During this re-examination, photographs, in combination with a comprehensive and standard clinical and digital examination will be taken. Further, patients will be given questionnaires to assess patient-reported outcomes. The evaluation visit will take place within a maximum of 1 hour, as the normal time required for a recall appointment on this type of patient with the presence of dental implants. Besides this one re-examination, no more visits will be necessary for the study outcomes. Data will be encrypted and collected in Redcap Software. The key for the encryption will be set up and stored by a person who is not involved in the study.

DETAILED DESCRIPTION:
Patients included in the previous case series study who received tooth replacement therapy with dental implants and maxillary sinus augmentation procedures will be invited for a recall exam at the Department of Oral Surgery to be part of this prospective case series study. During this recall exam, photographs, a comprehensive anamnesis, followed by a standard clinical and digital examination, as well as patient-reported outcomes will be performed.

Primary and secondary outcomes will be measured and collected, and it will be tested whether long-term MBL is smaller than the clinically relevant 5mm limit. As there is no reference group available and previously published raw data was presumably deleted due to data protection reasons, measurements of secondary outcomes will be summarized by calculating means (continuous data) or percentages (categorical data) including 95% confidence intervals, and compared to reported data from standard implant placement in other publications.

The reason for selecting this criterion is due to the new criteria published in the new classification of periodontal and peri-implant diseases and conditions, where a diagnosis of peri-implantitis should have 3mm of marginal bone levels respecting the implant's platform (Schwarz 2018).

To the best of the investigators' knowledge, this observational single-center study will be the first study providing the effectiveness of implant therapy in addition to sinus floor elevation procedures with a follow-up longer than 20 years. The findings of this study could bring a valuable perspective on the replacement of missing teeth with dental implants and could provide clinicians and researchers all over the world with reasons that guide the clinical decision-making process.

ELIGIBILITY:
Inclusion criteria:

* Patients who were initially treated at the Department of Oral Surgery and Stomatology between 1997 and 2001
* Implant placement in the presence of a sinus floor augmentation procedure received during this period
* Patients involved in a previous cohort study

Exclusion criteria will be patients:

* Not able to come to the re-examination
* Concomitant diseases that compromise the health of this subject during the comprehensive examination (i.e., active severe infectious diseases, liver or kidney dysfunction/failure, currently under treatment)
* Pregnant women, or unwilling to sign the consent form.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of interest will be recruited out of a cohort of patients who were initially treated at the Department of Oral Surgery and Stomatology between 1997 and 2001.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to assess the marginal bone loss (MBL) on the radiographs of implant-supported fixed partial dentures in patients who received maxillary sinus floor augmentation procedures. | 25 years
  Utilizing periapical radiographs

SECONDARY OUTCOMES:
Demographics | 25 years
  Age (years), sex, ethnicity, systemic factors, habits, oral hygiene techniques, frequency (times/day), and supportive periodontal/implant therapy (times/year).
Clinical parameters | 25 years
  Probing depth (mm), presence of bleeding on probing and suppuration on probing, gingival/mucosal recession (mm), keratinized tissue width (mm), mobility, mucosal thickness (mm), presence of local contributing factors (i.e., presence of aberrant frenum attachment).
Radiographic parameters | 25 years
  Marginal bone levels (mm), presence of periapical pathosis, distance from the adjacent teeth/implants (mm), presence of open contacts, efficacy of sinus augmentation procedure.
Implant-related | 25 years
  Length and dimension of the dental implant (mm), manufacturer, the timing of implant placement after extraction, needed for additional bone or soft tissue augmentation procedures.
Prosthetic-related | 25 years
  Analysis of occlusion (Dental-PreScale), integrity of prosthetic restoration (survival and success rates), technical complications, esthetic score (Pink and White Esthetic Scores), occlusal contacts.
Patient-reported Outcome Measures | 25 years
  Visual Analog Score for the use of Oral Health Impact Profile-14, Visual Analog Score for the satisfaction of the treatment, etc

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Couso-Queiruga, DDS, MS, Study Chair — University of Bern
Locations (1):
- School of Dental Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data will be provided in a further publication based on the cohort of patients and not by single individuals.